CLINICAL TRIAL: NCT00939900
Title: Multicenter, Open-labeled, Randomized Clinical Trial to Determine the Efficacy of Zoledronic Acid in Preventing Collapse of the Osteonecrotic Femoral Head
Brief Title: Efficacy of Zoledronic Acid in Preventing Collapse of the Osteonecrotic Femoral Head
Acronym: EZAPCOFH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Kyung-Hoi Koo, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HKR08T
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Avascular Necrosis of Femoral Head
Keywords: avascular necrosis of femoral head; bisphosphonate; collapse
MeSH Terms: conditions — Femur Head Necrosis; Unconsciousness | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aclasta (Experimental): aclasta group
  Interventions: Drug: zoledronic acid (aclasta)
- control (No Intervention): control group

INTERVENTIONS:
Drug: zoledronic acid (aclasta) — Once-yearly administration of 5mg zoledronic acid intravenously (dosage of treatment of osteoporosis) (+ calcium:1,200mg/day, VitD:800IU/day) during study period
  Other Names: aclasta
  Arms: aclasta

SUMMARY:
The purpose of this study is to test the effect of zoledronic acid over 2 years in preventing early collapse and progression of joint dome depression (≥ 2 mm by X-ray) of the femoral head in patients with large (> 30%: criteria according to Kim et al) nontraumatic osteonecrosis.

DETAILED DESCRIPTION:
Until now, the best treatment option in early (precollapse) large osteonecrosis femoral head is vascularizing fibular graft. However, it requires high microsurgical technique. Also it needs very long operation time (3-6hours), and morbidity associated with surgery is not low. In early stage osteonecrosis, osteoclasts are activated and resorb the necrotic portion of bone and osteoblasts are followed to lay down new bone. This process can weaken the bone function to support loading and can lead to collapse of bone. Bisphophonate can inhibit this osteoclastic bone resorption and enhance osteoblastic new bone formation. Recently, everyday oral intake of alendronate with vitamin D and calcium had a high success rate to prevent the collapse and decrease of hip joint pain in a short-term follow-up. However, the compliance or adherence to everyday oral intake is questionable. Moreover, the exact comparison based on MRI according to various classifications is not available currently. There is no report about the effect of zoledronic acid to prevent early collapse and progression of joint dome depression (≥2 mm by X-ray) of the early stage large nontraumatic osteonecrosis of the femoral head or its effect on MRI signal change after infusion of zoledronic acid in noncollapsed cases (estimated about 30% of cases) The investigators need a controlled randomized multicenter interventional study about the efficacy of bisphophonates in the treatment of ONFH.

ELIGIBILITY:
Inclusion Criteria:

* Patient who agree to clinical trial
* Patient who are more than 18 years of age
* Osteonecrosis of the femoral head
* Steinberg stage I, II non traumatic osteonecrosis of femoral head
* Necrotic area of > 30% (HJ Kim et al )
* JIC (Japanese Investigation Committee): C1 or C2 lateral lesion (by X-ray or MRI)

Exclusion Criteria:

* Patients who are pregnant (patients who are of child bearing potential who are not practicing a reliable contraceptive method (oral, subcutaneous, mechanical, or surgical contraception)
* Patients who have contraindicated condition to zoledronic acid such as chronic renal failure (calculated creatinine clearance less than 35.0 ml/min), severe heart disease such as atrial fibrillation, sensitive to bisphosphonates and hypocalcemia (serum calcium less than 8 mg/dl or 2.0 mmol/L)
* Patients who have collapsed lesion including subchonral fracture
* Patients who have multiple lesion of osteonecrosis of femoral head
* Patients who received other kinds of bisphophonates or anabolic agents before zoledronic acid use
* Patients with any medical or psychiatric condition which, in the Investigator's opinion would preclude the participant from adhering to the Protocol or completing the trial per protocol
* Patients who are considered potentially unreliable and patients who may not reliably attend study visits

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aclasta | Control
Started | 55 | 55
Completed | 53 | 48
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclasta | Control | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.8) | 45.2 (11.6) | 44.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Femoral Head Collapse Within 24 Months
Time Frame: Measurements were done at 6, 12, 24 months
Measure: Number; unit: participants
Arm/Group | Aclasta | Control
Number analyzed (Participants) | 53 | 48
participants | 29 | 22

2. Secondary Outcome: Collpase Rate of Femoral Head
Time Frame: Measurement will be done at 0m, 3m, 6m, 9m, 12m, 18m, 24m)
Reporting Status: Not Posted

3. Secondary Outcome: Change of HHS (Harris Hip Scores), WOMAC Score, SF-36
Time Frame: Measurement will be done at 0m, 3m, 6m, 9m, 12m, 18m, 24m)
Reporting Status: Not Posted

4. Secondary Outcome: Time to Collapse of Femoral Head
Time Frame: Measurement will be done at 0m, 3m, 6m, 9m, 12m, 18m, 24m)
Reporting Status: Not Posted

5. Secondary Outcome: Time to Total Arthroplasty or Joint Preserving Surgery
Time Frame: Measurement will be done at 0m, 3m, 6m, 9m, 12m, 18m, 24m)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aclasta | Control
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No